CLINICAL TRIAL: NCT02405884
Title: Effects of Hemodialysis on Intraocular Pressure in a University Hospital Located in Midwestern Brazil
Brief Title: Intraocular Pressure and Hemodialysis Midwestern Brazil
Acronym: EHPIOBRAZIL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VER Excelência em Oftalmologia (Other)
Responsible Party: Principal Investigator, Rodrigo Egidio da Silva, ophthalmologist, VER Excelência em Oftalmologia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20328813.0.0000.0037
Record Dates: First submitted 2015-03-24; First posted 2015-04-01 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-03

CONDITIONS: Renal Insufficiency, Chronic; Glaucoma
Keywords: Glaucoma; Renal Insufficiency, Chronic; Low Tension Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Renal Insufficiency, Chronic; Glaucoma; Low Tension Glaucoma; Ocular Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- measurement of intraocular pressure (Other): Patients were divided into groups according to the days on which they underwent hemodialysis. Intraocular pressure was measured with a Kowa HA-2 Perkins applanation tonometer. The tonometry included three measurements in the central region of the cornea before and after hemodialysis. In all patients, the measurements were performed three times on the days when hemodialysis sessions were performed, with 24 hours between each session, and the means of the measurements were obtained. All parameters were measured under prior corneal anesthesia with 0.1% proparacaine and 0.25% fluorescein eye drops.
  Interventions: Other: Kowa HA-2 Perkins applanation tonometer.

INTERVENTIONS:
Other: Kowa HA-2 Perkins applanation tonometer. — Patients were divided into groups according to the days on which they underwent hemodialysis. Intraocular pressure was measured with a Kowa HA-2 Perkins applanation tonometer. The tonometry included three measurements in the central region of the cornea before and after hemodialysis. In all patients, the measurements were performed three times on the days when hemodialysis sessions were performed, with 24 hours between each session, and the means of the measurements were obtained. All parameters were measured under prior corneal anesthesia with 0.1% proparacaine and 0.25% fluorescein eye drops.

SUMMARY:
Objective: To evaluate the variation in intraocular pressure in patients with chronic kidney disease, according to the time interval between hemodialysis sessions and to the influence of weight and blood pressure on intraocular pressure.

Methods: This was a cross-sectional study in which 78 eyes of 39 patients on hemodialysis, at the Santa Casa de Misericordia de Goiânia hospital, were analyzed in June 2014. Patients were divided into groups according to the days on which they underwent hemodialysis. The mean, standard deviation, and median of the intraocular pressure, blood pressure, and weight were calculated. P-values <0.05 were considered statistically significant.

DETAILED DESCRIPTION:
This cross-sectional observational study followed the guidelines of the Declaration of Helsinki, and all patients signed an informed consent form approved by the Ethics and Research Committee of the Pontifical Catholic University of Goiás (Pontifícia Universidade Católica de Goiás - PUC-GO). The inclusion criteria were chronic renal patients, who were older than 18 years of age, were part of the hemodialysis program of the Santa Casa de Misericordia de Goiânia (SCMG) hospital, signed the informed consent form and were able to undergo a physical examination. Exclusion criteria were patients on hemodialysis who were not chronic renal patients; patients who refused to participate in the study or could not undergo a physical examination; patients who did not undergo hemodialysis in the week of the study; prior ophthalmic eye disease or surgery; and patients allergic to anesthetic drops or dyes.

Patients were divided into groups according to the days on which they underwent hemodialysis. A total of 39 patients who were on hemodialysis at SCMG for six days in the month of June 2014 were analyzed. The patient's eye fundus was evaluated through direct ophthalmoscopy with a PanOptic device (Welch Allyn). Intraocular pressure was measured with a Kowa HA-2 Perkins applanation tonometer. The tonometry included three measurements in the central region of the cornea before and after hemodialysis. In all patients, the measurements were performed three times on the days when hemodialysis sessions were performed, with 24 hours between each session, and the means of the measurements were obtained. All parameters were measured under prior corneal anesthesia with 0.1% proparacaine and 0.25% fluorescein eye drops.

The variables studied were age, gender, base etiology for CKD, and variations in body weight and IOP before and after hemodialysis. Mean blood pressure (MBP), systolic blood pressure (SBP), diastolic blood pressure (DBP), and ocular perfusion pressure (OPP) were obtained before and after hemodialysis. The following mathematical models were used: MBP = (DBP) + 1/3 (SBP) - (DBP) and OPP = 2/3 (MBP-IOP), as described in the literature (18-20). The data were collected using a form devised for the study from the medical records of the chronic renal patients undergoing hemodialysis at SCMG and registered in the system.

The data were tabulated in a Microsoft© Excel 2007 spreadsheet and analyzed using the Statistical Package for the Social Sciences, version 20 (SPSS, Chicago, IL). The mean, standard deviation, median IOP measurements, blood pressure, and weight were obtained. Data normality was assessed by the Kolmogorov-Smirnov test. The significance of differences between measurements obtained before and after hemodialysis was assessed by the Wilcoxon test. The relationship between IOP and weight was assessed by Pearson's or Spearman's correlation. P-values <0.05 were considered significant.

ELIGIBILITY:
Inclusion Criteria:

* chronic renal patients
* Patientes signed the informed consent form and were able to undergo a physical examination
* Patients between 18-75 years of age

Exclusion Criteria:

* Patients with chronic eye disease and / or eye surgery
* Patients allergic to anesthetic drops or dyes.
* Patients who had no physical condition to the eye examination
* Patients who refused to participate in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2014-01; Primary Completion 2014-07 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
assess changes in intraocular pressure (mmHg) before and after hemodialysis | baseline (before hemodialysis ) and end of hemodialysis ( four hours late)

CONTACTS AND LOCATIONS:
Overall Officials: Francisco W Rodrigues, Professor, Principal Investigator — PUC Goias

REFERENCES:
- [Background] Hu J, Bui KM, Patel KH, Kim H, Arruda JA, Wilensky JT, Vajaranant TS. Effect of hemodialysis on intraocular pressure and ocular perfusion pressure. JAMA Ophthalmol. 2013 Dec;131(12):1525-31. doi: 10.1001/jamaophthalmol.2013.5599. PMID 24232671